CLINICAL TRIAL: NCT00731705
Title: In-Vitro Studies in Depletion of Haplotype Mismatched Alloreactive T Cells
Status: Withdrawn | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sherif Farag, MD, PhD, IU Simon Cancer Center
Organization: Indiana University (Other)
Other Study IDs: 0612-01/ IUCRO-0180
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Hematologic Malignancies; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood, apheresis samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients with hematological malignancies who are undergoing evaluation for autologous or allogeneic stem cell transplants OR First-degree relatives of patients evaluated for stem cell transplantation
  Interventions: Procedure: collection of peripheral blood and apheresis samples

INTERVENTIONS:
Procedure: collection of peripheral blood and apheresis samples — Sixty mL of peripheral blood will be collected from consenting eligible donors. Additionally, after the laboratory techniques have been fully evaluated, leukopheresis samples will also be collected.

SUMMARY:
The doctors in the Bone Marrow Transplant Service at the Indiana University Cancer Center are working to better understand how the immune cells that cause graft-versus-host disease (a major complication of stem cell transplantation in which the donor immune cells attack the patient's organs) can be selectively removed from the graft, leaving other immune cells that fight infections.

DETAILED DESCRIPTION:
The purpose of this research is to study how immune cells (called T cells) that cause graft-versus-host disease (GVHD) can best be selectively separated from other T cells and removed from the cells that will be returned to the cancer patient's body. These other T cells may protect against infection when given to patients after a stem cell transplant. The removal of cells that cause GVHD would allow doctors to safely give back the T cells that protect against infection, without the risk of GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies who are undergoing evaluation for autologous or allogeneic stem cell transplants will be eligible, if: (1)They have no circulating neoplastic cells in the peripheral blood as assessed by routine morphology or flow cytometry. (2)Patients with acute myeloid or lymphocytic leukemia are in complete remission
* First-degree relatives of patients evaluated for stem cell transplantation will be eligible if: (1) Willing to undergo testing for HIV and hepatitis B and C (free of charge) (2) Not pregnant at time of collection of blood (3)In good general health (4) No prior history of malignancy. (5) Age 18 years or older if donating apheresis product. (Because of the relatively invasive nature of the leukopheresis procedure and difficulties in obtaining consent, children <18 who are first degree relatives of the patient will not undergo apheresis for studies on this protocol)
* Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the Bone Marrow Transplant service at the Indiana University Melvin and Bren Simon Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
To develop the optimum conditions for activating the maximum number of alloreactive T cells from clinical scale samples | 5 years

SECONDARY OUTCOMES:
To develop a GMP grade high throughput, flow through immunomagnetic cell separation system for clinical scale depletion of alloreactive T cell, capable of t3log10 depletion of alloreactivity while retaining >80% third party reactivity. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center